CLINICAL TRIAL: NCT00824096
Title: Use Bronchoscopy to Predict Post-Extubation Stridor in Critical Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chimei Medical Center (Other)
Responsible Party: Kuo-Chen Cheng, Kuo-Chen Cheng
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CM-IRB09512014
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Post-Extubation Stridor
Keywords: endotracheal intubation; cuff-leak test; post-extubation stridor; bronchoscopy; corticosteroids; Cuff-leak volume less than 24%
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Bronchoscopy — The patients in our ICU intubated for > 24h and met weaning criteria, will be examined by bronchoscopy. Five ㏄ blood will be collected for checking CRP and cytokines before performing bronchoscopy. The proposed grading of post-extubation vocal cord finding were shown (Figure 1). The patients will be classified to two groups (Figure 2). The first group is these patients without swelling or swelling area ≦50% who will be extubated after bronchoscopic examination. These patients will be followed for 48 hours to monitor the incidence of PES. The second group is those patients who develop laryngeal edema with swelling area ≧50% or swelling in the whole vocal cord. Bosmin 2 ml local injection and Solu-medrol 40 mg I.V. Q6h for 1~4 days will be given. Bronchoscopy will be done if CLV ≧24% or after treatments for 3~4 days even with CLV <24%. The above treatments will be applied again if stridor develops. Extubation will be performed if no presence of laryngeal edema.

SUMMARY:
Our study aims at the accuracy of bronchoscopy to predict PES. Evidence base medicine guidelines for extubation may be obtained through this study.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater than 18 years old
* Intubation over 24 hrs
* Match weaning profile
* Cuff leak volume less than 24%
* VS and subject/family agree

Exclusion Criteria:

* Re-Intubation
* History of upper air way obstruction
* Severe CV disease (ex. AMI)
* Active UGI Bleeding
* Blood sugar persistent more than 250 mg/dl under medication control
* Risk of IICP
* Open T.B.
* Bleeding tendency/ Platelet less than 40 thousands
* Subject or family refuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The accuracy of bronchoscopy to predict post-extubation stridor. | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Intensive Care Medicine; Chi Mei Medical Center, Tainan, Taiwan